CLINICAL TRIAL: NCT05789823
Title: Efficacy and Safety of Ischemic Post-conditioning in Patients with Acute Ischemic Stroke After Mechanical Thrombectomy
Brief Title: Ischemic Post-conditioning in Acute Ischemic Stroke Thrombectomy (PROTECT-2)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROTECT-2
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Ischemic Postconditioning

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ischemic post-conditioning group (Experimental): Mechanical thrombectomy combined with ischemic post-conditioning
  Interventions: Procedure: Mechanical thrombectomy combined with ischemic post-conditioning
- Control group (Sham Comparator): Mechanical thrombectomy alone
  Interventions: Procedure: Mechanical thrombectomy alone

INTERVENTIONS:
Procedure: Mechanical thrombectomy combined with ischemic post-conditioning — Ischemic post-conditioning will be applied after successful recanalization of the culprit artery achieve by thrombectomy. Ischemic post-conditioning consists of briefly repeated 4 cycles × 2 minutes of occlusion and reperfusion (equal duration) of the initially occluded artery using a balloon.
  Arms: Ischemic post-conditioning group
Procedure: Mechanical thrombectomy alone — Successful recanalization was achieved by mechanical thrombectomy without subsequent ischemic post-conditioning.
  Arms: Control group

SUMMARY:
Ischemic post-conditioning is a neuroprotective strategy that has been proven to attenuate reperfusion injury in animal models of stroke. The investigators have conducted a 3 + 3 dose-escalation trial to demonstrate the safety and tolerability of ischemic post-conditioning incrementally for a longer duration of up to 5 min × 4 cycles in stroke patients undergoing mechanical thrombectomy. The purpose of this study is to further determine the efficacy and safety of ischemic post-conditioning in patients with acute ischemic stroke who are treated with mechanical thrombectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Acute ischemic stroke within 24 hours from stroke onset (or from time last known well) to groin puncture;
3. Previous mRS ≤ 2;
4. Baseline NIHSS ≥ 6;
5. Baseline ASPECTS ≥ 6;
6. Unilateral middle cerebral artery occlusion with or without ipsilateral internal carotid artery occlusion;
7. Successful recanalization after mechanical thrombectomy (eTICI 2b-3);
8. Written informed consent provided by the patients or their legal relatives.

Exclusion Criteria:

1. Confirmed or clinically suspected cerebral vasculitis/fibromuscular dysplasia;
2. Difficulty in reaching the designated position of the balloon used for ischemic post-conditioning;
3. Complications related to thrombectomy, such as contrast agent extravasation, vascular perforation/rupture, dissection, and escape of thrombus;
4. Stenting in the middle cerebral artery M1 segment/distal intracranial carotid artery during thrombectomy;
5. > 2 times of balloon dilations as rescue therapy due to angioplasty during thrombectomy;
6. Patients with contraindications to MRI;
7. Other conditions that the investigator considered inappropriate for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Infarct volume at 24 hours | 24 hours after randomization
  Infarct volume on MRI-DWI at 24 hours after randomization

SECONDARY OUTCOMES:
Progression of infarct volume between baseline and 24 hours | Baseline and 24 hours after randomization
  Difference of infarct volume on MRI-DWI between baseline and 24 hours after randomization
Progression of perfusion defect from baseline to 24 hours | Baseline and 24 hours after randomization
  The volume difference of Tmax > 6 s from baseline to 24 hours after randomization
Progression of infarct volume between 2 hours and 24 hours | 2 hours after randomization and 24 hours after randomization
  Difference of infarct volume on MRI-DWI between 2 h after randomization and 24 h after randomization
Infarct volume at 5 days/at discharge | 5 days after randomization or at discharge
  Infarct volume on CT/MRI-FLAIR at 5 days after randomization/at discharge
The proportion of functional independence at 90 days | 90 days after randomization
  The modified Rankin Scale (mRS) score of 0-2 at 90 days after randomization; the mRS is an ordinal disability score of 7 categories (0=no symptoms to 5=severe disability, and 6=death)
The proportion of favorable outcome at 90 days | 90 days after randomization
  The mRS score of 0-3 at 90 days after randomization; the mRS is an ordinal disability score of 7 categories (0=no symptoms to 5=severe disability, and 6=death)
The distribution of mRS score at 90 days | 90 days after randomization
  The distribution of the mRS score at 90 days after randomization; the mRS is an ordinal disability score of 7 categories (0=no symptoms to 5=severe disability, and 6=death)
National Institute of Health Stroke Scale (NIHSS) score at 24 hours | 24 hours after randomization
  NIHSS score at 24 hours after randomization; the NIHSS ranges from 0 to 42, with higher scores indicating more severe neurologic deficits
The proportion of early neurological improvement | Baseline and 24 hours after randomization
  NIHSS 0-2 or ≥ 8 lower than baseline NIHSS score at 24 hours after randomization; the NIHSS ranges from 0 to 42, with higher scores indicating more severe neurologic deficits
National Institute of Health Stroke Scale (NIHSS) score at 5 days/at discharge | 5 days after randomization or at discharge
  NIHSS score at 5 days after randomization/at discharge; the NIHSS ranges from 0 to 42, with higher scores indicating more severe neurologic deficits
Recanalization rate at 24 hours | 24 hours after randomization
  Recanalization rate at 24 hours after randomization (eTICI 2b-3)
Cerebral blood flow velocity of the culprit middle cerebral artery at 24 hours after randomization. | 24 hours after randomization
  Cerebral blood flow will be assessed by transcranial Doppler ultrasound at 24 hours after randomization

OTHER OUTCOMES:
Safety outcome (mortality at 90 days) | 90 days after randomization
  90-day mortality
Safety outcome (the proportion of symptomatic intracranial hemorrhage within 24 hours) | Within 24 hours after randomization
  The proportion of symptomatic intracranial hemorrhage within 24 hours after randomization
Safety outcome (the proportion of intracranial hemorrhage within 24 hours) | Within 24 hours after randomization
  The proportion of intracranial hemorrhage within 24 hours after randomization
Safety outcome (the proportion of malignant brain edema within 24 hours) | Within 24 hours after randomization
  The proportion of malignant brain edema within 24 hours after randomization
Procedure-related complications | During the procedure
  Vascular perforation/rupture, vessel dissection, severe vasospasm, rupture of the balloon used for post-conditioning

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Huanhu Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Wu L, Wei M, Zhang B, Zhang B, Chen J, Wang S, Luo L, Liu S, Li S, Ren C, Hess DC, Song H, Zhao W, Ji X. Safety and Tolerability of Direct Ischemic Postconditioning Following Thrombectomy for Acute Ischemic Stroke. Stroke. 2023 Sep;54(9):2442-2445. doi: 10.1161/STROKEAHA.123.044060. Epub 2023 Jul 27. PMID 37497674
- [Background] Wu L, Zhang B, Zhao W, Ji X, Wei M. Ischemic post-conditioning in acute ischemic stroke thrombectomy: A phase-I duration escalation study. Front Neurosci. 2022 Dec 8;16:1054823. doi: 10.3389/fnins.2022.1054823. eCollection 2022. PMID 36523440
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/36523440/